CLINICAL TRIAL: NCT05562115
Title: Proteomic Study of Tears From Patients With a PAX6 Mutation
Acronym: PLAPAX6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL22_0050
Record Dates: First submitted 2022-09-21; First posted 2022-09-30 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Aniridia
Keywords: PAX6; tear proteomics; aniridia
MeSH Terms: conditions — Aniridia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients treated for an ocular malformation linked to a PAX6 mutation. (Experimental)
  Interventions: Other: Tear collection

INTERVENTIONS:
Other: Tear collection — Collection of tears by Schirmer strip (2 to 4 mm).

SUMMARY:
This is a single-center prospective pilot study involving the ophthalmology and medical genetics departments of the Montpellier University Hospital, and the proteomics platform of the Montpellier University Hospital.

5 patients with PAX6 pathogenic variation will be included in order to determine the proteomic profile in a tear sample associated with different pathogenic variations of the PAX6 gene.

Participation in the study for the patients consists of a single visit with an ophthalmological examination and a tear collection.

DETAILED DESCRIPTION:
The transcription factor PAX6 is required for the normal development of all elements constituting the eyeball, including the lacrimal gland.

In patients with PAX6 gene mutations, the cornea presents a limbal anomaly that has been evolving since childhood and is responsible for variable damage. It evolves from a simple peripheral keratopathy to an advanced stage with complete corneal opacification and fibrosis. Chronic inflammation, associated with tear film damage is very common and promotes keratopathy. The current treatment of dry eye in patients with ocular malformation related to a PAX6 mutation is non specific: it aims to palliate the quantitative tear defect and uses tear substitutes, cyclosporine eye drops, meatus plugs, scleral lenses.

The identification of specific qualitative abnormalities constitutes the indispensable preliminary step necessary in order to be able to consider in the long term an adapted treatment, of tear protein supplementation, aiming at preserving the cornea of patients with an ocular malformation related to a PAX6 gene mutation.

In this study, patients will be recruited from the active file of patients and patients previously treated in the ophthalmology or medical genetics departments of Montpellier University Hospital for an ocular malformation related to a PAX6 mutation.

Participation in the study will consist of a single visit of up to 3 hours.

During the pre-inclusion visit, the existence of a pathogenic variation of the PAX6 gene identified in each patient will be verified.

Once the inclusion is achieved, the same day, it is planned to:

* data collection: demographic (age, sex), clinical (weight, height, head circumference, blood pressure, associated neurodevelopmental disorder, neurological examination, extraocular damage, description of the ocular malformation, previous surgical interventions) and genetic (description of the pathogenic variation of the PAX6 gene),
* an ophthalmological examination,
* the collection of tears by Schirmer strip (2 to 4 mm) will be performed by the ophthalmologist.

The data for each protein in the spectrum will be compared with the previously established reference proteomic profile range. Significant variations (50% change) will be retained.

The discovery of tear film abnormalities in the pathophysiological context of a PAX6 gene alteration will allow a better understanding of the progressive tear and corneal damage in these complex ocular malformations. This is an essential preliminary step in the perspective of a better management of the patients, by the creation of specific adapted eye drops allowing to palliate more specifically the identified anomalies, following the example of the treatment by eye drops containing NGF developed in the United States in order to treat the attacks of the corneal innervation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with an isolated pathogenic variation of PAX6
2. Age: 18-60 years
3. Subject affiliated to a French social security system or beneficiary of such a system
4. Written consent given by the subject

Exclusion Criteria:

1. Ophthalmologic procedure less than 3 months old
2. Chromosomal abnormality not limited to the PAX6 gene
3. Being under court protection, guardianship or curatorship
4. To be deprived of liberty by administrative decision
5. Be in a period of exclusion in relation to another protocol
6. Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
Proteomic profile of tears associated with different pathogenic variations of the PAX6 gene. | Through study completion, an average of 18 months
  Proteomic profile (quantitative and qualitative analysis of global protein expression after gel prefractionation) of tears associated with different pathogenic variations of the PAX6 gene.

SECONDARY OUTCOMES:
Types of changes relative to the previously established reference tear profile range. | Through study completion, an average of 18 months
  Types of changes (protein expression deficiency or excess, defined as greater than 50% change) relative to the previously established reference tear profile range.

CONTACTS AND LOCATIONS:
Overall Officials: Marjolaine WILLEMS, PH, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital, Montpellier, France